CLINICAL TRIAL: NCT03744910
Title: A Pivotal Phase 3 Trial to Evaluate the Safety and Efficacy of Clazakizumab for the Treatment of Chronic Active Antibody-mediated Rejection in Kidney Transplant Recipients
Brief Title: Clazakizumab for the Treatment of Chronic Active Antibody Mediated Rejection in Kidney Transplant Recipients
Acronym: IMAGINE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early stop for lack of efficacy/futility (at Interim analysis)
Sponsor: CSL Behring (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL300_3001; 2018-003682-34 (EudraCT Number); VKTX01 (Other: Vitaeris)
Record Dates: First submitted 2018-11-06; First posted 2018-11-19 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Antibody-mediated Rejection
Keywords: Chronic Active; Antibody-mediated Rejection (AMR)
MeSH Terms: interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazakizumab (Active Comparator): Clazakizumab is a genetically engineered humanized immunoglobulin G1 (IgG1) mAb that binds to human IL-6 that is administered subcutaneously.
  Interventions: Biological: Clazakizumab
- Placebo (Placebo Comparator): Physiologic saline solution that is administered subcutaneously.
  Interventions: Drug: Physiologic saline solution

INTERVENTIONS:
Biological: Clazakizumab — Clazakizumab is a genetically engineered humanized immunoglobulin G1 (IgG1) mAb that binds to human IL-6
  Arms: Clazakizumab
Drug: Physiologic saline solution — Normal saline
  Arms: Placebo

SUMMARY:
This trial investigates the efficacy and safety of clazakizumab [an anti-interleukin (IL)-6 monoclonal antibody (mAb)] for the treatment of CABMR in recipients of a kidney transplant.

ELIGIBILITY:
* Inclusion criteria:

  1. Age 18-75 years.
  2. Living donor/deceased donor kidney transplant recipients ≥6 months from time of transplant.
  3. Diagnosis of CABMR determined by kidney biopsy and the presence of HLA DSA using single-antigen bead-based assays. For eligibility, kidney biopsy must not be older than 12 months and DSA analysis must be performed no longer than 6 months prior to the start of Screening.

     NOTE: • Within 3 months prior to the start of Screening, treatments for ABMR or TCMR, with the exception of steroids*, are not allowed (see Exclusion Criterion 3).

     • If treatment for ABMR (including CABMR) or TCMR (other than steroids*) was given between 3 to 12 months of Screening, a repeat kidney biopsy and DSA analysis are required at least 6 weeks after the end of treatment to confirm continuing CABMR and presence of HLA DSA and to determine eligibility.

     * A maximum dose of 2g of methylprednisolone intravenously (or dose equivalent of other steroids), followed by a taper to the original maintenance steroid dose is allowed.

     The following histopathologic and serologic diagnostic criteria (based on Banff 2015 criteria [Loupy et al, 2017]) must be met for inclusion:
     1. Morphologic evidence of chronic tissue injury, as demonstrated by transplant glomerulopathy (TG) (cg) > 0). Biopsies without evidence of chronic tissue injury on light microscopy, but with glomerular basement membrane double contours on electron microscopy (cg1a) are eligible.
     2. Evidence of current/recent antibody interaction with vascular endothelium, including 1 or more of the following:

     i. Linear C4d staining in peritubular capillaries or medullary vasa recta (Banff scores C4d2 or C4d3 by immunofluorescence on frozen sections, or C4d > 0 by immunohistochemistry on paraffin sections).

     ii. At least moderate microvascular inflammation ([glomerulitis score, g + peritubular capillaritis score, ptc] ≥ 2) in the absence of recurrent or de novo glomerulonephritis, although in the presence of acute TCMR, borderline infiltrate, or infection, ptc ≥ 2 alone is not sufficient and g must be ≥ 1.

     NOTE: The local pathologist's diagnosis must be reviewed by a central pathologist to confirm eligibility for entry into the study. Biopsies with other histopathologic changes (eg, BKV nephropathy or recurrent glomerulonephritis) may be eligible if concurrent CABMR changes (as detailed above) are present and determined to be the predominant cause of renal dysfunction.

     c. Serologic evidence of circulating HLA DSA. NOTE: The local laboratory DSA results must be reviewed and confirmed by the central HLA reviewer during the screening period.
  4. Written informed consent obtained from subject (or legally acceptable representative) before any trial-related procedures.
* Exclusion criteria:

  1. Multi-organ transplant recipient (except for simultaneous kidney-pancreas or previous multiple kidney transplants) or cell transplant (islet, bone marrow, stem cell) recipient.
  2. Treatment for ABMR (including CABMR) or TCMR within 3 months prior to the start of screening with the exception of steroids.
  3. Received T cell depleting agents (e.g., alemtuzumab, anti-thymocyte globulin) within 3 months prior to the start of screening.
  4. Pregnant, breastfeeding, or unwillingness to practice adequate contraception.
  5. Active tuberculosis (TB) or history of active TB.
  6. History of human immunodeficiency virus (HIV) infection or positive for HIV.
  7. Seropositive for hepatitis B surface antigen (HBsAg)
  8. Hepatitis C virus (HCV) RNA positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (141):
- United States (49):
  - University of Alabama at Birmingham (UAB) - University of Alabama Hospital (UAB Hospital), Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Keck Medical Center Of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Kidney Transplant Research Program, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - California Institute of Renal Research, San Diego, California
  - North America Research Institute, San Dimas, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - University Of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Tampa General Medical Group, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center - University Cardiovascular Surgeons, Chicago, Illinois
  - Indiana University (IU) Health Physicians - Kidney Diseases Clinic - Medical Diagnostic Center Location, Indianapolis, Indiana
  - Unity Point Health, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Massachusetts General Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine - Infectious Diseases (WU ID) Clinic, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center Corp., Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - New York Presbyterian Hospital / Weill Cornell Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Comprehensive Transplant Center, Columbus, Ohio
  - University of Cincinnati, Toledo, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Central Pennsylvania Transplant Foundation, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Renal Disease Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - VCU Health, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health (UWSMPH), Madison, Wisconsin
  - Medical College of WI Froedtert Hospital, Milwaukee, Wisconsin
- Australia (13):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - WSLHD, Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The University of Queensland - Princess Alexandra Hospital (PAH), Woolloongabba, Queensland
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital (SCGH), Nedlands, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton
  - Linear Clinical Research, Nedlands
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - LKH-Universität Hospital Graz, Graz
  - Universitätsklinik für Innere Medizin III Innsbruck, Innsbruck
  - Medizinische Universität Wien, Allgemeines Krankenhaus der S, Vienna
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- Canada (10):
  - Vancouver General Hospital - Gordon & Leslie Diamond Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Providence Health Care, Univ. Of British Columbia, Vancouver, British Columbia
  - Shared Health Inc. operating as the Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Health Centre, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - St Paul's Hospital Foundation, Saskatoon, Saskatchewan
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal (CRCHUM), Montreal
  - University Health Network, Toronto
- Czechia (3):
  - Centrum kardiovaskulární a transplantacní chirurgie Brno, Brno-střed
  - Fakultní Nemocnice Olomouc, Olomouc
  - IKEM, Prague
- France (17):
  - CHU GRENOBLE ALPES - Consultation Néphrologie Bureau des ARC (Côté Chartreuse, Rez-de-Chaussée Haut), Grenoble, Grenoble Cédex 09
  - Néphrologie - Pavillon Sainte Venise - CHU de Rouen - Hôpital de Bois Guillaume, Bois-Guillaume
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire (CHU) - Hopital Henri Mondor, Créteil
  - Hopital Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire (CHU) De Limoges Hopital Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital de la Conception - APHM, Marseille
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier Arnaud de Villeneuve, Montpellier
  - CHU de Nantes - Houtel Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice, Hopital Pasteur 2, Nice
  - Hospital Saint-Louis - APHP, Paris
  - Hopital Necker Enfants Malades, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hopitaux Universitaire de Strasbourg-Centre de References des Maladies Autoimmunes, Strasbourg
  - CHU Rangueil, Toulouse
  - Centre Hospitalier Regional Universitaire de Tours (CHRU de Tours) - Hopital Bretonneau, Tours
- Charite - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin, Germany
- Hungary (2):
  - Debreceni Egyetem, Klinikai Központ, Auguszta, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Netherlands (8):
  - Amsterdam University Medical Center (Amsterdam UMC), Academic Medical Center (AMC), Amsterdam
  - Amsterdam UMC location AMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht University Medical Centre, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Auckland City Hospital, Auckland, New Zealand
- South Korea (13):
  - Pusan National University Hospital, Busan
  - Keimyung Dongsan Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kosin University Gospel Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (10):
  - Hospital Del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre-Centro de Actividades Ambulatorias, Madrid
  - Hospital Universitario Marques De Valdecilla, Santander
  - Centro Hospital Universitario Dr. Preset, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Karolinska University Hospital, Huddinge
  - Karolinska University Hospital, Solna
  - Uppsala Universitet - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Hualien City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichang
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

REFERENCES:
- [Derived] Mannon RB, Vincenti FG. Poised for Innovation: Considerations for End Points for New Drug Development in Kidney Transplantation. J Am Soc Nephrol. 2024 Nov 1;35(11):1603-1606. doi: 10.1681/ASN.0000000000000475. Epub 2024 Aug 5. No abstract available. PMID 39102302
- [Derived] Nickerson PW, Bohmig GA, Chadban S, Kumar D, Mannon RB, van Gelder T, Lee JC, Adler S, Chong E, Djamali A. Clazakizumab for the treatment of chronic active antibody-mediated rejection (AMR) in kidney transplant recipients: Phase 3 IMAGINE study rationale and design. Trials. 2022 Dec 22;23(1):1042. doi: 10.1186/s13063-022-06897-3. PMID 36550562
- [Derived] Borski A, Eskandary F, Haindl S, Doberer K, Muhlbacher J, Mayer KA, Budde K, Halloran PF, Chong E, Jilma B, Bohmig GA, Wahrmann M. Anti-interleukin-6 Antibody Clazakizumab in Antibody-mediated Renal Allograft Rejection: Accumulation of Antibody-neutralized Interleukin-6 Without Signs of Proinflammatory Rebound Phenomena. Transplantation. 2023 Feb 1;107(2):495-503. doi: 10.1097/TP.0000000000004285. Epub 2023 Jan 26. PMID 35969004
- [Derived] Jordan SC, Ammerman N, Choi J, Huang E, Najjar R, Peng A, Sethi S, Sandhu R, Atienza J, Toyoda M, Ge S, Lim K, Gillespie M, Zhang X, Haas M, Vo A. Evaluation of Clazakizumab (Anti-Interleukin-6) in Patients With Treatment-Resistant Chronic Active Antibody-Mediated Rejection of Kidney Allografts. Kidney Int Rep. 2022 Feb 9;7(4):720-731. doi: 10.1016/j.ekir.2022.01.1074. eCollection 2022 Apr. PMID 35497778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 139 study sites in 13 countries: Canada, United States, Austria, Czechia, France, Germany, Hungary, Netherlands, Spain, Sweden, Switzerland, Democratic People's Republic of Korea, and Australia.
Pre-assignment Details: A total of 382 participants were screened, of which 188 were screen failures. Of the screened participants, 194 were randomized in a 1:1 ratio to receive study interventions (Clazakizumab or Placebo).
Groups:
- Clazakizumab: Participants received clazakizumab via subcutaneous (SC) injection once every 4 weeks (Q4W) until the participant: permanently discontinued the investigational product (IP), withdrew from the study, experienced allograft loss, died, or reached the common treatment end date (CTED), whichever occurred first during this study.
- Placebo: Participants received Placebo by SC injection Q4W until the participant: permanently discontinued IP, withdrew from the study, experienced allograft loss, died, or reached the CTED, whichever occurred first during this study.
Period: Overall Study
Arm/Group | Clazakizumab | Placebo
Started | 94 | 100
Completed (Participants that reached the primary endpoint of allograft loss or death.) | 16 | 15
Not Completed | 78 | 85
Not completed — Withdrew Consent | 1 | 8
Not completed — Physician Decision | 5 | 4
Not completed — Sponsor Decision (due to study termination) | 68 | 71
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other-unspecified | 4 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized set, which included all participants who were randomized.
Groups:
- Clazakizumab: Participants received clazakizumab via SC injection Q4W until the participant: permanently discontinued the IP, withdrew from the study, experienced allograft loss, died, or reached the CTED, whichever occurred first during this study.
- Placebo: Participants received Placebo via SC injection Q4W until the participant: permanently discontinued IP, withdrew from the study, experienced allograft loss, died, or reached the CTED, whichever occurred first during this study.
- Total: Total of all reporting groups
Arm/Group | Clazakizumab | Placebo | Total
Number analyzed (Participants) | 94 | 100 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.87) | 47.0 (12.24) | 46.7 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 65 | 74 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic, Latino/a or of Spanish origin | 69 | 78 | 147
  Ethnicity: Hispanic, Latino/a or of Spanish origin | 18 | 16 | 34
  Ethnicity: Not reported | 5 | 4 | 9
  Ethnicity: Unknown | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 62 | 69 | 131
  Race: Black or African American | 10 | 7 | 17
  Race: Korean | 9 | 13 | 22
  Race: Other | 6 | 8 | 14
  Race: Asian Indian | 3 | 1 | 4
  Race: Other Asian | 2 | 1 | 3
  Race: American or Alaskan Native | 1 | 0 | 1
  Race: Filipino | 1 | 0 | 1
  Race: Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 52 in Estimated Glomerular Filtration Rate (eGFR)
Description: This primary outcome measure was the one from the first interim analysis.
Time Frame: From Baseline to Week 52
Population: Analysis was performed on the intent-to-treat (ITT) analysis set. The ITT analysis set consisted of all randomized participants who received at least 1 dose of study drug and who had a baseline assessment and at least 1 post baseline assessment of eGFR.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per minute per 1.73 meter^2
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
milliliter per minute per 1.73 meter^2 | -8.0 [-10.2 to -5.8] | -5.2 [-7.4 to -3.1]
Statistical Analysis 1: Comparison: Clazakizumab vs Placebo; Test type: Other; Treatment difference = -2.75, 95% CI 2-sided [-5.84 to 0.35], Standard Error of Mean 1.563

2. Primary Outcome: Number of Participants With Composite All-cause Allograft Loss or Irreversible Loss of Allograft Function
Description: Composite all-cause allograft loss or irreversible loss of allograft function, defined as time to first occurrence of any of the following components:
  * eGFR < 15 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2)*
  * return to dialysis*
  * allograft nephrectomy
  * retransplantation
  * death from any cause, or
  * a sustained (greater than or equal to [>=] 60 days) 40% decline in eGFR from Baseline.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.)
  If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The number of participants with composite all-cause allograft loss or irreversible loss of allograft function are reported here. Time-to-event data were not calculated due to the study's termination.
Time Frame: From Baseline to 4 years
Population: Analysis was performed on the ITT analysis set. The ITT analysis set consisted of all participants who received at least 1 dose of study drug and who had a baseline assessment and at least 1 post baseline assessment of eGFR.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 26 | 22

3. Primary Outcome: Percentage of Participants With Composite All-cause Allograft Loss or Irreversible Loss of Allograft Function
Description: Composite all-cause allograft loss or irreversible loss of allograft function, defined as time to first occurrence of any of the following components:
  * eGFR < 15 mL/min/1.73 m^2*
  * return to dialysis*
  * allograft nephrectomy
  * retransplantation
  * death from any cause, or
  * a sustained (greater than or equal to [>=] 60 days) 40% decline in eGFR from Baseline.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.)
  If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The percentage of participants with composite all-cause allograft loss or irreversible loss of allograft function are reported here.
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
percentage of participants | 28.3 | 22.2

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and Adverse Events of Special Interest (AESIs)
Time Frame: Up to 4 years
Population: Analysis was performed on the safety analysis set (SAS). The SAS consisted of all randomized participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 100
Participants
  TEAEs | 89 | 88
  Serious TEAEs | 39 | 39
  AESIs | 56 | 52

5. Primary Outcome: Percentage of Participants With TEAEs, Serious TEAEs, and AESIs
Time Frame: Up to 4 years
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 100
percentage of participants
  TEAEs | 95.7 | 88.0
  Serious TEAEs | 41.9 | 39.0
  AESIs | 60.2 | 52.0

6. Primary Outcome: Number of Participants Who Tested Positive for Polyoma BK Virus (BKV), Cytomegalovirus (CMV) and Epstein-Barr Virus (EBV)
Description: Number of participants who tested positive for BKV, CMV or EBV according to the maximum measured viral amount (International Units/mL [IU/mL]) after baseline are reported here.
Time Frame: From baseline up to 4 years
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 100
Participants
  BKV >Lower limit of quantification (LLOQ) to <320 IU/mL: number analyzed (Participants) | 93 | 99
  BKV >Lower limit of quantification (LLOQ) to <320 IU/mL | 3 | 2
  BKV >=320 IU/mL to <3200 IU/mL: number analyzed (Participants) | 93 | 99
  BKV >=320 IU/mL to <3200 IU/mL | 1 | 0
  BKV >=3200 IU/mL: number analyzed (Participants) | 93 | 99
  BKV >=3200 IU/mL | 1 | 0
  CMV >LLOQ to <1000 IU/mL: number analyzed (Participants) | 93 | 99
  CMV >LLOQ to <1000 IU/mL | 5 | 1
  CMV >=1000 IU/mL to <5000 IU/mL: number analyzed (Participants) | 93 | 99
  CMV >=1000 IU/mL to <5000 IU/mL | 2 | 2
  CMV >=5000 IU/mL: number analyzed (Participants) | 93 | 99
  CMV >=5000 IU/mL | 0 | 0
  EBV >LLOQ to <10200 IU/mL: number analyzed (Participants) | 92 | 99
  EBV >LLOQ to <10200 IU/mL | 8 | 7
  EBV >=10200 IU/mL to <20400 IU/mL: number analyzed (Participants) | 92 | 99
  EBV >=10200 IU/mL to <20400 IU/mL | 0 | 0
  EBV >=20400 IU/mL: number analyzed (Participants) | 92 | 99
  EBV >=20400 IU/mL | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Laboratory Test Results
Description: Laboratory tests included liver function test (LFTs), complete blood count (CBC), plasma lipids, high-sensitivity C-reactive protein (hsCRP). Only participants with abnormal laboratory test results are reported here. Here, ULN = upper limit of normal, LLN = lower limit of normal, ALT = Alanine aminotransferase and AST = Aspartate aminotransferase.
Time Frame: Up to 4 years
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug. Here, 'overall number of participants analyzed' = participants with evaluable data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 99
Participants
  ALT : >ULN to 3 x ULN | 15 | 6
  ALT : > 3 to 5 × ULN | 0 | 1
  AST : >ULN to 3 x ULN | 11 | 4
  AST : > 3 to 5 × ULN | 1 | 0
  AST : > 5 × ULN | 0 | 2
  Bilirubin: > ULN to 2 × ULN | 20 | 6
  Bilirubin: > 2 × ULN | 5 | 0
  Neutrophils: < 2.5 to 1.5 10^9/L | 33 | 21
  Neutrophils: < 1.5 to 1.0 10^9/L | 15 | 5
  Neutrophils: < 1.0 10^9/L | 7 | 0
  Platelets: < LLN to 75.0 10^9/L | 39 | 10
  Platelets: < 75.0 to 50.0 10^9/L | 1 | 0

8. Primary Outcome: Percentage of Participants With Abnormal Laboratory Test Results
Description: Laboratory tests included LFTs, CBC, plasma lipids, hsCRP. Only percentage of participants with abnormal laboratory test results are reported here. Here, ULN = upper limit of normal, LLN = lower limit of normal, ALT = Alanine aminotransferase and AST = Aspartate aminotransferase.
Time Frame: Up to 4 years
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 99
percentage of participants
  ALT : >ULN to 3 x ULN | 16.1 | 6.1
  ALT : > 3 to 5 × ULN | 0 | 1.0
  AST : >ULN to 3 x ULN | 11.8 | 4.0
  AST : > 3 to 5 × ULN | 1.1 | 0
  AST : > 5 × ULN | 0 | 2.0
  Bilirubin: > ULN to 2 × ULN | 21.5 | 6.1
  Bilirubin: > 2 × ULN | 5.4 | 0
  Neutrophils: < 2.5 to 1.5 10^9/L | 35.5 | 21.2
  Neutrophils: < 1.5 to 1.0 10^9/L | 16.1 | 5.1
  Neutrophils: < 1.0 10^9/L | 7.5 | 0
  Platelets: < LLN to 75.0 10^9/L | 41.9 | 10.1
  Platelets: < 75.0 to 50.0 10^9/L | 1.1 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Change in Vital Signs, Electrocardiograms (ECGs), and Physical Examination
Time Frame: Up to 4 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 100
Participants | 0 | 0

10. Primary Outcome: Number of Participants With Positive Anti-drug Antibodies
Time Frame: Baseline, Weeks 12, 24, and 48
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug. Here, 'overall number of participants' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 88 | 97
Participants
  Baseline | 5 | 10
  Week 12: number analyzed (Participants) | 74 | 82
  Week 12 | 3 | 8
  Week 24: number analyzed (Participants) | 68 | 72
  Week 24 | 2 | 7
  Week 48: number analyzed (Participants) | 52 | 52
  Week 48 | 0 | 4

11. Primary Outcome: Percentage of Participants With Positive Anti-drug Antibodies
Time Frame: Baseline, Weeks 12, 24, and 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 88 | 97
percentage of participants
  Baseline | 5.7 | 10.3
  Week 12: number analyzed (Participants) | 74 | 82
  Week 12 | 4.1 | 9.8
  Week 24: number analyzed (Participants) | 68 | 72
  Week 24 | 2.9 | 9.7
  Week 48: number analyzed (Participants) | 52 | 52
  Week 48 | 0 | 7.7

12. Secondary Outcome: Number of Participants With Composite All-cause Allograft Loss
Description: Composite all-cause allograft loss, defined as, time to first occurrence of any of the following components:
  * eGFR < 15 mL/min/1.73 m^2*
  * return to dialysis*
  * allograft nephrectomy
  * retransplantation, or
  * death from any cause.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.) If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The number of participants with composite all-cause allograft loss are reported here.
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 17 | 14

13. Secondary Outcome: Percentage of Participants With Composite All-cause Allograft Loss
Description: Composite all-cause allograft loss, defined as, time to first occurrence of any of the following components:
  * eGFR < 15 mL/min/1.73 m^2*
  * return to dialysis*
  * allograft nephrectomy
  * retransplantation, or
  * death from any cause.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.) If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The percentage of participants with composite all-cause allograft loss are reported here.
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
percentage of participants | 18.5 | 14.1

14. Secondary Outcome: Number of Participants With Irreversible Loss of Allograft Function
Description: Irreversible loss of allograft function as defined by a 40% decline in eGFR from Baseline sustained for at least 60 days.
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 22 | 18

15. Secondary Outcome: Percentage of Participants With Irreversible Loss of Allograft Function
Description: as for outcome 14
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
percentage of participants | 23.9 | 18.2

16. Secondary Outcome: Number of Participants With Death-censored Allograft Loss
Description: Time to death-censored allograft loss, was defined as occurrence of any of the following components:
  * eGFR < 15 mL/min/1.73 m^2*
  * return to dialysis*
  * allograft nephrectomy, or
  * retransplantation.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.) If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The number of participants with death-censored allograft loss are reported here.
Time Frame: From Baseline to 4 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 16 | 13

17. Secondary Outcome: Percentage of Participants With Death-censored Allograft Loss
Description: Death-censored allograft loss was defined as the occurrence of any of the following components:
  * eGFR < 15 mL/min/1.73 m^2*
  * return to dialysis*
  * allograft nephrectomy, or
  * retransplantation.
  (*Total cumulative duration of sustained eGFR < 15 mL/min/1.73 m^2 AND / OR dialysis >= 60 days.)
  If the eGFR < 15 mL/min/1.73 m^2 was the only component reached, the value must be sustained over at least 60 days and must be confirmed by a repeat measurement after >= 60 days from the first measurement. The percentage of participants who experienced death-censored allograft loss are reported here.
Time Frame: From Baseline to 4 years
Population: Analysis was performed on the ITT analysis set. The ITT analysis set consisted of all randomized participants who received at least 1 dose of the investigational product, had a Baseline assessment, and had at least 1 post-baseline assessment of eGFR.
Measure: Number; unit: percentage of participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
percentage of participants | 17.4 | 13.1

18. Secondary Outcome: Change From Baseline in Urine Albumin Creatinine Ratio (UACR)
Time Frame: From Baseline to Week 52
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: gram per mole
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 83 | 88
gram per mole | 50.734 (125.5628) | 31.178 (112.8894)

19. Secondary Outcome: Percent Change From Baseline in Mean Fluorescent Intensity for Donor-Specific Antibodies (DSA)
Time Frame: From Baseline to Week 52
Population: Analysis was performed on the SAS. The SAS consisted of all randomized participants who had received at least 1 dose of study drug. The Overall Number of Participants Analyzed reported here reflects all participants who were analyzed, which includes all (N = 93 Clazakizumab and 100 Placebo) participants assessed at baseline to determine DSA class I or II. Here, 'Number Analyzed' = the number of participants in Class I or II classified at baseline who had available MFI data at Week 52.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 93 | 100
percent change
  DSA Class I: number analyzed (Participants) | 21 | 16
  DSA Class I | -23.20 [-53.34 to -4.54] | -39.71 [-69.67 to -20.22]
  DSA Class II: number analyzed (Participants) | 39 | 45
  DSA Class II | -27.15 [-46.32 to -5.05] | -13.68 [-26.69 to -1.75]

20. Secondary Outcome: Change From Baseline in Banff Lesion Grading Score (2015 Criteria) of Pre-treatment to Post-treatment (Week 52) Kidney Biopsies
Description: Banff lesion grading scores assess the presence and the degree of histopathological changes in the different compartments of kidney biopsies. Here, the improved category is defined as a decline in the Banff lesion grading score. Participants with improved scores, not improved scores, and missing biopsies for C4d staining, interstitial fibrosis, tubular atrophy, glomerular basement membrane double contours, glomerulitis and peritubular capillaritis are reported for this outcome measure.
Time Frame: From Baseline to Week 52
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants
  C4d Staining: Improved score | 10 | 10
  C4d Staining: Not improved score | 17 | 21
  C4d Staining: Missing biopsies | 65 | 68
  Interstitial Fibrosis: Improved score | 3 | 8
  Interstitial Fibrosis: Not improved score | 24 | 23
  Interstitial Fibrosis: Missing biopsies | 65 | 68
  Tubular Atrophy: Improved score | 1 | 5
  Tubular Atrophy: Not improved score | 26 | 26
  Tubular Atrophy: Missing biopsies | 65 | 68
  Glomerular Basement Membrane Double Contours: Improved score | 6 | 10
  Glomerular Basement Membrane Double Contours: Not improved score | 21 | 21
  Glomerular Basement Membrane Double Contours: Missing biopsies | 65 | 68
  Glomerulitis: Improved score | 14 | 17
  Glomerulitis: Not improved score | 13 | 14
  Glomerulitis: Missing biopsies | 65 | 68
  Peritubular Capillaritis: Improved score | 14 | 15
  Peritubular Capillaritis: Not improved score | 13 | 16
  Peritubular Capillaritis: Missing biopsies | 65 | 68

21. Secondary Outcome: Incidence of Acute Rejection Episodes of T Cell-mediated Rejection (TCMR) and Antibody-mediated Rejection (ABMR)
Description: Number of participants who had at least one acute rejection episode (TCMR or ABMR) are reported for this outcome measure.
Time Frame: Baseline up to End of treatment (up to approximately 4 years)
Population: Analysis was performed on the ITT analysis set. The ITT analysis set consisted of all randomized participants who received at least 1 dose of study drug and who had a baseline assessment and at least 1 post baseline assessment of eGFR.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 2 | 3

22. Secondary Outcome: Overall Participant Survival
Description: Number of participants who were alive up to Week 52 are reported for this outcome measure.
Time Frame: Up to Week 52
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 92 | 99
Participants | 90 | 98

23. Secondary Outcome: Maximum Concentration at Steady State (Cmax ss) of CSL300
Description: A subset of participants (out of the enrolled participants in the main study) had the option to participate in a pharmacokinetic (PK)/ Pharmacodynamic (PD) sub-study.
Time Frame: Up to Week 24
Population: Analysis was performed on the PK/ PD analysis set. The PK/PD substudy analysis set consisted of all participants in the SAS who consented to be a part of the PK / PD substudy and had at least 1 quantifiable PK concentration of investigational product after administration. Here, "overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Clazakizumab
Number analyzed (Participants) | 3
nanograms per milliliter | 3556.8 (10.5)

24. Secondary Outcome: Trough Concentrations at Steady State (Ctrough ss) of CSL300
Description: A subset of participants (out of the enrolled participants in the main study) had the option to participate in a PK/PD sub-study.
Time Frame: Up to Week 24
Population: Analysis was performed on the PK/PD analysis set. The PK/PD substudy analysis set consisted of all participants in the SAS who consented to be a part of the PK / PD substudy and had at least 1 quantifiable PK concentration of investigational product after administration. Here, "overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Clazakizumab
Number analyzed (Participants) | 3
nanograms per milliliter | 2366.8 (9.2)

25. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-tau) at Steady State of CSL300
Description: as for outcome 24
Time Frame: Up to Week 24
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*nanograms per milliliter
Arm/Group | Clazakizumab
Number analyzed (Participants) | 3
days*nanograms per milliliter | 78080.34636 (7.19614)

26. Secondary Outcome: Time of Maximum Concentration at Steady State (Tmax ss) of CSL300
Description: as for outcome 24
Time Frame: Up to Week 24
Population: as for outcome 24
Measure: Median (Full Range); unit: day
Arm/Group | Clazakizumab
Number analyzed (Participants) | 3
day | 6.92292 [4.9986 to 11.9299]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: The SAS consisted of all randomized participants who received at least 1 dose of study drug. The participants in the SAS were analyzed according to the actual treatment received.
Arm/Group | Clazakizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/93 | 1/100
Serious Adverse Events (participants affected / at risk) | 39/93 | 39/100
Other Adverse Events (participants affected / at risk) | 81/93 | 80/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (N=93) | Placebo (N=100)
COVID-19 (Infections and infestations) | 13 (15) | 10 (12)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephriti (Infections and infestations) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 13 (15) | 6 (7)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (3)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complications of transplanted pancreas (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Lymphatic obstruction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 2 (2)
Chronic allograft nephropathy (Immune system disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (3) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Renal and pancreas transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (N=93) | Placebo (N=100)
COVID-19 (Infections and infestations) | 28 (31) | 30 (31)
Urinary tract infection (Infections and infestations) | 12 (21) | 6 (9)
Nasopharyngitis (Infections and infestations) | 5 (6) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 5 (6)
Herpes zoster (Infections and infestations) | 6 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 21 (24) | 22 (25)
Nausea (Gastrointestinal disorders) | 11 (13) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 7 (7)
Vomiting (Gastrointestinal disorders) | 10 (12) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (14) | 13 (18)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 16 (19) | 16 (17)
Neutropenia (Blood and lymphatic system disorders) | 15 (22) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 8 (14) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8) | 1 (1)
Oedema peripheral (General disorders) | 24 (31) | 11 (12)
Fatigue (General disorders) | 8 (9) | 8 (10)
Asthenia (General disorders) | 1 (1) | 5 (5)
Blood creatinine increased (Investigations) | 9 (12) | 13 (15)
Immunosuppressant drug level decreased (Investigations) | 4 (9) | 6 (10)
Immunosuppressant drug level increased (Investigations) | 4 (6) | 6 (10)
Weight decreased (Investigations) | 3 (3) | 6 (6)
Blood bilirubin increased (Investigations) | 5 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 5 (5)
Proteinuria (Renal and urinary disorders) | 5 (5) | 8 (8)
Renal impairment (Renal and urinary disorders) | 7 (7) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 8 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 12 (12) | 13 (15)
Headache (Nervous system disorders) | 10 (14) | 9 (9)
Insomnia (Psychiatric disorders) | 6 (7) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was not able to complete secondary endpoint assessments as planned. The study was terminated due to futility after the planned interim analysis based on the change in eGFR from baseline to Week 52 and analysis was conducted where feasible using the data collected at Week 52 or by the time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03744910/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03744910/SAP_001.pdf